CLINICAL TRIAL: NCT05845476
Title: Sexual Orientation and Gender Identity (SOGI) Data Collection Program Implementation and Evaluation
Acronym: SOGI
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Arthur, Principal Investor, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-22301
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Cancer Surveillance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SOGI Data Collection Intervention: This single arm is an educational intervention for clinicians. After consent, they provide baseline survey fata, then the training intervention, then a post assessment.
  Interventions: Other: Patient SOGI Self-Report; Other: SOGI Resource for Clinical Care Education (SORCE); Other: Cancer Center Care Environment

INTERVENTIONS:
Other: Patient SOGI Self-Report — EPIC® MyChart electronic health records messages will go to OSUCCC patients of pilot clinics who have incomplete SOGI data in their record and are enrolled in OSU MyChart. The message will request that patients complete SOGI data fields, with an explanation about why it is important for their health care, as well as links to document this information in their electronic health record (EHR).
  Intervention Description:
  EPIC® MyChart EHR messages will go to OSUCCC patients of pilot clinics who have incomplete SOGI data in their record and are enrolled in OSU MyChart. The message will request that patients complete SOGI data fields, with an explanation about why it is important for their health care, as well as links to document this information in their electronic health record.
Other: SOGI Resource for Clinical Care Education (SORCE) — SOGI Resource for Clinical Care Education (SORCE) training includes cultural competency and health education. SORCE training has been used on a smaller scale for two years at the OSUCCC-James, receiving excellent scores for presentation quality, knowledge gained, and presenter expertise. For the present study, SORCE training will be tailored based on results from Aim 1. The training curriculum includes didactic content (basics of the LGBTQ+ community, SOGI data collection for patient care and research, and social determinants of health for the LGBT community, 15 minutes), EHR SOGI data documentation demonstration (10 minutes), and open dialogue and role play (20 minutes). Trainees will be given EHR documentation tip sheets and laminated pocket cards with best practices for asking about SOGI, steps for documenting in the EHR, and additional resources.
Other: Cancer Center Care Environment — At the level of the OSUCCC, to include all inpatient and ambulatory spaces, the investigators will implement important measures aimed at changing culture and practice. This includes modification of policy and the EHR for SOGI documentation per National Academy of Science Engineering and Medicine recommendations, a multi-pronged approach to making the environment of care more visibly welcoming for SGM people, and leveraging existing diversity, equity, and inclusion structures and initiatives to shift culture at the cancer center.

SUMMARY:
Sexual and gender minority (SGM) individuals experience significant cancer-related health disparities across the cancer continuum. The overall goal of this proposal is to assess multi-level barriers associated with sexual orientation and gender identity (SOGI) data collection in the health record as well as implementation factors including feasibility, acceptability, and data completeness. The results of this study will make a significant impact by making SOGI data available for research, addressing barriers to SOGI data collection in a large comprehensive cancer center, and informing compassionate cancer care for SGM people.

DETAILED DESCRIPTION:
Sex and gender minority people (SGM, i.e., lesbian, gay, bisexual, transgender, queer, and other people of diverse sexual orientation or gender identity (SOGI) experience significant cancer-related health disparities across the cancer continuum. SGM people have an increased risk for some cancers, may be diagnosed at more advanced stages of the disease, and have poor mental health outcomes. Despite calls from national organizations for systematic collection of SOGI data, this information is not routinely collected in health research or clinical health records, perpetuating the invisibility of SGM people in research and clinical care and fueling health disparities. Systematic and standardized collection of SOGI data is necessary for assessing cancer-related health outcomes through cancer registries, for comparing outcomes and care delivery in clinical trials, and for providing culturally relevant care for SGM people. Barriers to systematic SOGI data collection come from patient, clinician, and system levels. Multilevel barriers to SOGI data collection require a multilevel approach to create standardized, systematic program implementation and evaluation at cancer centers across the country. Barriers and best practices for SOGI data collection likely differ by region and institutional history and culture. Ohio is traditionally a conservative 'red' state, with large rural and Appalachian regions. The catchment area for The Ohio State University Comprehensive Cancer Center (OSUCCC) encompasses Ohio's 88 counties and nearly 11.8 million people -- many of whom come from diverse, and often underserved, populations including urban, rural, Appalachia, immigrant, Amish, and SGM communities. Thus, OSUCCC is well-positioned to make a significant impact in the health of SGM Ohioans through systematic SOGI data collection and improved SGM-sensitive clinical care and culture. The overall goal of this Administrative Supplement is to assess multi-level barriers associated with SOGI data collection as well as implementation factors including feasibility, acceptability, and data completeness. To accomplish this goal, the investigators propose two aims. First, the investigators will develop effective strategies to collect SOGI data based on barriers and facilitators identified at the patient, staff/provider, and cancer center levels. The investigators will accomplish this through community and patient focus groups, staff/provider interviews, and a cancer center environmental scan. Second, the investigators will implement a systematic SOGI data collection program at the patient, staff/provider, and cancer center levels with systematic program evaluation at all levels. The investigators will accomplish this through patient self-report, staff/provider training, and changes in cancer center medical record, policy, and environment of care. This proposal is innovative because our SOGI data collection program operates at multiple levels within the healthcare delivery context and includes both central medical campuses and satellite clinics. The results of this study will make a significant impact by 1) making SOGI data available for cancer registries, 2) addressing factors associated with implementation in a large comprehensive cancer center, and 3) informing culturally responsive cancer care for SGM Ohioans.

ELIGIBILITY:
Inclusion Criteria:

Aim 1

* Community group members that represent sex and gender minority (SGM) people
* Cisgender/ heterosexual patients and family members
* Ambulatory clinic provider and staff responsible for collecting sexual orientation and gender identity (SOGI) data
* Age ≥18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Able to provide informed consent
* Able to read and speak English

Aim 2

* Ambulatory clinic providers and staff responsible for collecting sexual orientation and gender identity (SOGI) data
* Age ≥18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Able to provide informed consent
* Able to read and speak English

Exclusion Criteria

1. Language or technology barriers that limit data collection
2. Insufficient evidence of meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * SGM community groups and OSUCCC-James patient advocacy group for feedback on best practices from collecting SOGI data
  * OSUWMC Staff/Faculty: Recruit faculty and staff through the directories at the 3 pilot test clinic sites (thoracic clinic, breast-surgical oncology clinic, and hematology lymphoma clinic) to integrate SOGI data collection into clinical workflows. Faculty and staff will be recruited via meeting announcements and emails.
  Participants will be JPAS and clinical staff from ambulatory departments at the 3 pilot clinics responsible for collecting SOGI data from OSUCCC-James patients. Ambulatory faculty and staff responsible for SOGI data collection will be systematically trained and begin data collection as part of their routine job responsibilities.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Sexual Orientation Documentation | Baseline (prior to intervention)
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Sexual Orientation Documentation | 1 month post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Sexual Orientation Documentation | 2 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Sexual Orientation Documentation | 3 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Sexual Orientation Documentation | 4 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Sexual Orientation Documentation | 5 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Sexual Orientation Documentation | 6 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with sexual orientation documented), percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | Baseline (prior to intervention)
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | 1 month post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | 2 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | 3 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | 4 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | 5 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Gender Identity Documentation | 6 months post intervention
  This variable is observed from the electronic health record (EHR) and reported in aggregate form. The investigators will record and analyze the count (number of patients with gender identity documented percent of patient records containing this documentation out of the total number of patient records, and completeness of variable fields (count and percent).
Clinics with Staff/Provider Training Completed | Baseline (prior to intervention)
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.
Clinics with Staff/Provider Training Completed | 1 month post intervention
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.
Clinics with Staff/Provider Training Completed | 2 months post intervention
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.
Clinics with Staff/Provider Training Completed | 3 months post intervention
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.
Clinics with Staff/Provider Training Completed | 4 months post intervention
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.
Clinics with Staff/Provider Training Completed | 5 months post intervention
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.
Clinics with Staff/Provider Training Completed | 6 months post intervention
  The investigators will record and analyze the count (number of staff, providers, and clinics that have completed the tailored cultural competency and EHR documentation training; SORCE) as well as the percent of staff, providers, and clinics trained out of the total number selected for training and program implementation.

SECONDARY OUTCOMES:
Staff and Provider Implementation Survey | Baseline (prior to intervention)
  The investigators will administer a brief, online survey of trained staff and clinicians evaluating awareness or comfort level with SOGI data collection, workflow integration, and obstacles to implementation.
Staff and Provider Implementation Survey | Immediately post intervention
  The investigators will administer a brief, online survey of trained staff and clinicians evaluating awareness or comfort level with SOGI data collection, workflow integration, and obstacles to implementation.
Staff and Provider Implementation Survey | Month 6 post intervention
  The investigators will administer a brief, online survey of trained staff and clinicians evaluating awareness or comfort level with SOGI data collection, workflow integration, and obstacles to implementation.
Patient Experience Data | Baseline (prior to intervention)
  OSUCCC Patient Experience department provides data on patient concerns (presented at point of care) and complaints (formal and written complaints) by type and frequency. Concerns and complaints specifically related to SOGI data collection or the care of SGM people will be reported.
Patient Experience Data | 3 months post intervention
  OSUCCC Patient Experience department provides data on patient concerns (presented at point of care) and complaints (formal and written complaints) by type and frequency. Concerns and complaints specifically related to SOGI data collection or the care of SGM people will be reported.
Patient Experience Data | 6 months post intervention
  OSUCCC Patient Experience department provides data on patient concerns (presented at point of care) and complaints (formal and written complaints) by type and frequency. Concerns and complaints specifically related to SOGI data collection or the care of SGM people will be reported.
Environmental Scan Checklist | Baseline (prior to intervention)
  Environmental scan checklist includes chart reviews, review of internal documents (e.g. intake forms) and policies, and assessment of the physical environment (e.g. gendered colors or names, presence of gender-neutral restroom, rainbow flag or other sign of safety, gendered waiting rooms) by study staff for identification of the ways the physical and virtual spaces may be unwelcoming to or discriminatory against SGM people
Environmental Scan Checklist | 6 months post intervention
  Environmental scan checklist includes chart reviews, review of internal documents (e.g. intake forms) and policies, and assessment of the physical environment (e.g. gendered colors or names, presence of gender-neutral restroom, rainbow flag or other sign of safety, gendered waiting rooms) by study staff for identification of the ways the physical and virtual spaces may be unwelcoming to or discriminatory against SGM people
Clinical Cancer-Related Outcomes | 12-month project completion
  From the electronic health record, The investigators will obtain cancer-related health outcome data for SGM people and matched controls (cisgender, heterosexual people) to include vital status, cancer stage and recurrence, second cancers, and mental and physical functioning.
  From the electronic health record, The investigators will obtain cancer-related health outcome data for SGM people and matched controls (cisgender, heterosexual people) to include vital status, cancer stage and recurrence, second cancers, and mental and physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Arthur, PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The James Line — http://cancer.osu.edu